CLINICAL TRIAL: NCT05190614
Title: Radiographic Evaluation of a Star-shaped Incision Technique for Thick-gingiva and Thin-gingiva Patients Treated With Implant-supported Fixed Prosthesis: a Randomized Trial
Brief Title: Radiographic Evaluation of a Star-shaped Incision Technique
Status: Completed | Type: Observational
Sponsor: Wen Luo (Other)
Responsible Party: Sponsor-Investigator, Wen Luo, Associate Professor, West China Hospital
Organization: West China Hospital (Other)
Other Study IDs: 2019021
Record Dates: First submitted 2021-12-14; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Clinical and Radiographic Effect; Thick-gingiva; Thin-gingiva; Implant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- thick-gingiva group: After the insertion of the probe into the facial aspect of the sulcus through the gingival margin, the simple visual method is based on the transparency of the periodontal probe through the gingival margin while probing the buccal sulcus at the midfacial aspect of the tooth. When the outline of the underlying periodontal probe can't be seen through the gingival, the gingival phenotype is considered thick.
- thin-gingiva group: After the insertion of the probe into the facial aspect of the sulcus through the gingival margin, the simple visual method is based on the transparency of the periodontal probe through the gingival margin while probing the buccal sulcus at the midfacial aspect of the tooth. When the outline of the underlying periodontal probe can be seen through the gingival, the gingival phenotype is considered thin.
  Interventions: Diagnostic Test: The biotype of gingiva

INTERVENTIONS:
Diagnostic Test: The biotype of gingiva — The biotype of gingival was determined by periodontal probe.
  Groups: thin-gingiva group

SUMMARY:
To evaluate a star-shaped incision technique to thick-gingiva and thingingiva patients treated with implant-supported fixed prosthesis. The star-shaped incision would be an effective and simple method to reconstruct gingival papillae and avoid the gingival recession in thick-gingiva patients treated with implant-supported fixed prosthesis, and it is worthy of clinical extend.

DETAILED DESCRIPTION:
Objective: To evaluate a star-shaped incision technique to thick-gingiva and thin-gingiva patients treated with implant-supported fixed prosthesis. Methods and Materials: 24 patients received cross-shaped incision were assigned into thick-gingiva group (16 cases) and thin-gingiva group (8 cases). Follow-up examination was carried out 3 and 12 months after final restoration. Clinical and radiographic evaluation including gingival papilla height, modified plaque index, modified sulcus bleeding index, periodontal depth, and crestal marginal bone level were utilized.

ELIGIBILITY:
Inclusion criteria

1. Good general health, no chronic systemic diseases.
2. All subjects included in this study needed to have one missing premolar or molar teeth with adjacent natural teeth.
3. All subjects included in this study had been treated with one bone-level implant insertion in the premolar or molar region. The patients had insufficient gingival papilla height (referred to contralateral natural tooth which also had insufficient gingival papilla height) and at least 2 mm of keratinized tissue width around the implant.

Exclusion criteria

1. Active periodontal infections.
2. Heavy smoking (> 10 cigarettes per day).

Ages: 22 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study samples were comprised of patients who had been treated with one bone-level implant (Osstem, Korea) insertion in the premolar or molar region. Twenty-four subjects were selected from the patients who came to the Department of Oral Implantology, West China Hospital of Stomatology, Sichuan University in China between June 2019 and June 2021.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Papilla height | Between June 2019 and June 2021
  Presence/absence of papilla height was assessed visually according to the papilla index proposed by Jemt
Modified Plaque Index (mPI) | Between June 2019 and June 2021
  plaque accumulation around the marginal peri-implant tissue was assessed by the criteria of mPI
Modified Sulcus Bleeding Index (mBI) | Between June 2019 and June 2021
  the bleeding tendency of the marginal peri-implant tissue was evaluated using mBI
Probing Depth (PD, mm) | Between June 2019 and June 2021
  PD was assessed at the mid-buccal, mid-oral, mesial and distal aspects of the buccal surfaces of each implant with a standard periodontal probe, and final value was determined by the average of four aspects.
Gingival margin level (GML) | Between June 2019 and June 2021
  gingival margin level was assessed by calculating the vertical distance between the most apical point of gingival margin at the buccal aspect of the crown and line connecting the peak of the adjacent mesial and distal natural teeth (PMD)
The landmarks of first bone-implant contact (fBIC) and implant shoulder (IS) | Between June 2019 and June 2021
  fBIC-IS was defined as the vertical distance the first bone-implant contact to implant shoulder, and the distance was assessed at the mesial and distal aspect of implant, respectively. When the marginal crestal bone was located coronal to the IS, a positive (+) value was given, where a negative (-) value when located apically to the IS, the value was deemed as zero when IS and fBIC coincided. The crestal bone level at the time of impression taking was regarded as baseline. The known implant length was used for the calibration of dimensional distortion in the radiograph (the length of implant was 10 mm).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Zheng, MD, Principal Investigator — West China Hospital of Stomatology, Sichuan University, China
Locations (1):
- West China Hospital of Stomatology, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Du H, Gao M, Qi C, Liu S, Lin Y. Drug-induced gingival hyperplasia and scaffolds: they may be valuable for horizontal food impaction. Med Hypotheses 2010;74(6): 984-5. 2. Bidra AS. Nonsurgical management of inflammatory periimplant disease caused by food impaction: a clinical report. J Prosthet Dent 2014;111(2): 96-100. 3. Berglundh T, Lindhe J, Ericsson I, Mainello CP, Lijenberg B. The soft tissue barrier at implants and teeth. Clin Oral Implants Res 1991; 2: 81-90. 4. Berglundh T, Lindhe J, Jonsson K, Ericsson I. The topography of the vascular systems in the periodontal and peri-implant tissues in the dog. J Clin Periodontol 1994; 21: 189-93. 5. Chow YC, Wang HL. Factors and techniques influencing peri-implant papillae. Implant Dent 2010; 19(3): 208-19. 6. Sanavi F, Weisgold AS, Rose LF. Biologic width and its relation to periodontal biotypes. J Esthet Dent 1998; 10(3): 157-63. 7. De Rouck T, Eghbali R, Collys K, De Bruyn H, Cosyn J. The gingival biotype revisited: transparency of the periodontal probe through the gingival margin as a method to discriminate thin from thick gingiva. J Clin Periodontol 2009; 36(5): 428-33. 8. Olsson M, Lindhe J. Periodontal characteristics in individuals with varying form of the upper central incisors. J Clin Periodontol 1991; 18(1): 78-82. 9. Pontoriero R, Carnevale G. Surgical crown lengthening: a 12-month clinical wound healing study. J Periodontol 2001;72(7): 841-8. 10. Ronay V, Sahrmann P, Bindl A, Attin T, Schmidlin PR. Current status and perspectives of mucogingival soft tissue measurement methods. J Esthet Restor Dent 2011; 23(3):146-56. 11. Mombelli A, van Oosten MA, Schurch E Jr, Land NP. The microbiota associated with successful or failing osseointegrated titanium implants. Oral Microbiol Immunol 1987; 2(4):145-51. 12. Chang M, Wenstrom JL, Odman P, Andersson B. Implant supported single-tooth replacements compared to contralateral natural teeth. Crown and soft tissue dimensions. Clin Oral Implants Res 1999; 10(3): 185-94. 13. Welander M, Abrahamsson I, Berglundh T. The mucosal barrier at implant abutments of different materials. Clin Oral Implants Res 2008;19(7): 635-41. 14. Kajiwara N, Masaki C, Mukaibo T, Kondo Y, Nakamoto T, Hosokawa R. Soft tissue biological response to zirconia and metal implant abutments compared with natural tooth: microcirculation monitoring as a novel bioindicator. Implant Dent 2015; 24(1): 37-41. 15. Muller HP, Heinecke A, Schaller N, Eger T. Masticatory mucosa in subjects with different periodontal phenotypes. J Clin Periodontol 2000; 27(9):621-6. 16. Pradeep AR, Karthikeyan BV. Peri-implant papilla reconstruction: realities and limitations. J Periodontol, 2006. 77(3): p. 534-44. 17. Kan JY, Rungcharassaeng K, Umezu K, Kois JC. Dimensions of peri-implant mucosa: an evaluation of maxillary anterior single implants in humans. J Periodontol 2003;74(4):557-62. 18. Finelle G, Papadimitriou DE, Souza AB, Katebi N, Gallucci GO, Araujo MG. Peri-implant soft tissue and marginal bone adaptation on implant with non-matching healing abutments: micro-CT analysis. Clin Oral Implants Res, 2015; 26(4): e42-6. 19. Farronato D, Santoro G, Canullo L, Botticelli D, Maiorana C, Lang NP. Establishment of the epithelial attachment and connective tissue adaptation to implants installed under the concept of
- [Derived] Luo W, Kuang H, Sun H, Huang Y, Wang J, Zheng K, Li Z, Qu Y, Man Y, Wu Y. Star-shaped incision technique for gingiva patients treated with implant-supported fixed prosthesis. Medicine (Baltimore). 2023 Jul 7;102(27):e34324. doi: 10.1097/MD.0000000000034324. PMID 37417601